CLINICAL TRIAL: NCT01932775
Title: An Open, Single-centre, Non-controlled Study of Efficacy, Safety and Usability of the GlucoTab System for Glycaemic Management in Non-critically Ill Patients With Type 2 Diabetes at General Wards
Brief Title: Efficacy, Usability Study of the GlucoTab System for Glycaemic Management in Type 2 Diabetic Patients at General Wards
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ClinDiab-04
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GlucoTab System (Experimental)
  Interventions: Device: GlucoTab System

INTERVENTIONS:
Device: GlucoTab System

SUMMARY:
Objective: To investigate the performance (safety) of the GlucoTab system for glycaemic management in non-critically ill patients with type 2 diabetes at general wards.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged ≥18 years
* Type 2 diabetes (treated with diet, oral agents, non-insulin injected anti-diabetic medicine, insulin therapy or any combination of the four) or newly diagnosed hyperglycaemia which requires s.c. insulin therapy

Exclusion Criteria:

* Type 1 diabetes, gestational diabetes
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient
* Pregnancy
* Any mental condition rendering the patient incapable of giving his consent
* Known or suspected allergy to insulin glargine or insulin aspart
* Continuous parenteral nutrition
* Participation in another trial which can influence the software algorithm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mean percentage of blood glucose measurements in the target range 70 to 140 mg/dl, as calculated by all premeal and bedtime glucose values measured ≥ 24 hours after start of therapy | duration of hospital stay (maximum three weeks)

SECONDARY OUTCOMES:
Number of blood glucose measurements per day | duration of hospital stay (maximum three weeks)
Adherence to the insulin dose suggestion of the GlucoTab system | duration of hospital stay (maximum three weeks)
Mean daily blood glucose as calculated by premeal and bedtime blood glucose values: Overall and per treatment day | duration of hospital stay (maximum three weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University of Graz, Department of Internal Medicine, Division of Endocrinology and Metabolism
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Donsa K, Beck P, Holl B, Mader JK, Schaupp L, Plank J, Neubauer KM, Baumgartner C, Pieber TR. Impact of errors in paper-based and computerized diabetes management with decision support for hospitalized patients with type 2 diabetes. A post-hoc analysis of a before and after study. Int J Med Inform. 2016 Jun;90:58-67. doi: 10.1016/j.ijmedinf.2016.03.007. Epub 2016 Mar 23. PMID 27103198
- [Derived] Schaupp L, Donsa K, Neubauer KM, Mader JK, Aberer F, Holl B, Spat S, Augustin T, Beck P, Pieber TR, Plank J. Taking a Closer Look--Continuous Glucose Monitoring in Non-Critically Ill Hospitalized Patients with Type 2 Diabetes Mellitus Under Basal-Bolus Insulin Therapy. Diabetes Technol Ther. 2015 Sep;17(9):611-8. doi: 10.1089/dia.2014.0343. Epub 2015 Apr 30. PMID 25927357